CLINICAL TRIAL: NCT05898880
Title: The Effect of Self-Administered Acupressure and Acupressure Applied by Therapist on Pain, Nausea-Vomiting, and Mental Well-Being in Oncology Patients: A Three-Arm Randomized Controlled Study
Brief Title: The Effect of Acupressure on Pain, Nausea-Vomiting, and Mental Well-Being in Oncology Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Esra Cavusoglu, Principal Investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: mERSİNuU.
Record Dates: First submitted 2023-05-22; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Pain; Nausea With Vomiting Chemotherapy-Induced; Mental Health Wellness 1
Keywords: Chemotherapy; Pain; Nausea-vomiting; Mental Well-Being; Acupressure
MeSH Terms: conditions — Pain; Psychological Well-Being | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This is a prospective, three-armed (1:1:1), randomized controlled experimental single-blind clinical trial.
Who Masked: Investigator
Masking Description: Patients included in the study will not be blinded as they will be in acupressure (administered by the therapist), self-acupressure or control groups.
  Researchers will be blinded only during group assignment. The data will be transferred to the computer environment by the researchers, and a biostatistician independent of the research will analyze the data and report the findings without knowing which of the three groups are. Thus, the biostatistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self acupressure group (Experimental): The first acupressure application will be administered and taught individually by the researcher to the oncology patients in the self-administered group. Afterwards, each patient who learns the application will be asked to apply acupressure on his own for three days. In the self-acupressure group, a questionnaire form consisting of a personal information form, visual analog scale, nausea, vomiting and retching index and mental well-being scale will be applied first (pre-test) before the acupressure application is taught to the group by the researchers. Afterwards, patients will apply acupressure on their own for three days, and at the end of this period (post-test), a questionnaire consisting of personal information form, visual analog scale, nausea, vomiting and retching index and mental well-being scale will be applied. Acupressure will be applied the large intestine meridian 4th Point (LI4), the pericardium meridian Neiguan (P6) and Yintang (EX-HN3).
  Interventions: Other: Self-acupressure
- Acupressure by therapist (Other): In this group, acupressure will be administered to stage I, stage II, and stage III cancer patients receiving at least one course of chemotherapy for a total of three days by researchers with acupressure certification. Before the application (pre-test) by the therapist, a questionnaire consisting of a personal information form, visual analog scale, nausea, vomiting and retching index and mental well-being scale will be applied to the patients in the group in question. At the end of the three-day acupressure application (post-test) applied to the patients included in the study by the therapist, a questionnaire consisting of a personal information form, visual analog scale, nausea, vomiting and retching index and mental well-being scale will be applied. In the acupressure group applied by the therapist, a total of three points will be applied to the upper extremity: the 4th point of the large intestine meridian (LI4), the Pericardium Meridian/Neiguan (P6), Yintang (EX-HN3) point.
  Interventions: Other: Acupressure by therapists
- Control group (Other): The control group will receive the routine treatment applied in the hospital, and acupressure will not be applied to this group.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Self-acupressure — In the self-acupressure group, before the application, the tissue sensitivity will be reduced by heating and rubbing for 20 seconds without direct pressure on the acupressure points, and the points will be made ready for acupressure application. Afterwards, sequential (breathing rhythm) compressions will be applied to the determined acupressure points by the researcher for a total of two minutes for each point without raising the finger, taking into account the pain threshold of the individual who is applied with the thumb, with 10 seconds of pressure for two seconds of relief. Two of the three different points (LI4 and P6) selected for the application will be applied symmetrically on the other extremity. Therefore, the session duration of each patient will be approximately 12 minutes, depending on the preparation and compression time on each point. Afterwards, acupressure will be applied to themselves by participants
  Arms: Self acupressure group
Other: Acupressure by therapists — In the acupressure group applied by therapist, before the application, the tissue sensitivity will be reduced by heating and rubbing for about 20 seconds without direct pressure on the acupressure points, and the points will be ready for acupressure application. Afterwards, sequential (breathing rhythm) compressions will be applied to the determined acupressure points by the researcher for a total of two minutes for each point without raising the finger, taking into account the pain threshold of the individual who is applied with the thumb, with 10 seconds of pressure for two seconds of relief. Two of the three different points (LI4 and P6) selected for the application will be applied symmetrically on the other extremity. Therefore, the session duration of each patient will be approximately 12 minutes, depending on the preparation and compression time on each point.
  Arms: Acupressure by therapist
Other: Control group — No intervention will be made in the control group.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to compare the effect of self acupressure and acupressure applied by therapists on pain, nausea-vomiting, and mental well-being in oncology patients.

For this purpose, 93 individuals with stage 1-stage 3 cancer will be included in the study.

The main questions it aims to answer are:

• Is acupressure effective on pain, nausea-vomiting and mental well-being in oncology patients? Is there a difference in the effectiveness of self-acupressure and acupressure applied by therapist on pain, nausea-vomiting and mental well-being? The participants will be included in the study as three groups, namely the self-acupressure group, the acupressure group applied by the therapist, and the control group.

Self-acupressure participants will self-administer acupressure. In the acupressure group, which will be applied by the therapist, acupressure will be applied to the participants by researchers who have acupressure certificate.

In the control group, acupressure etc. No additional application will be made. Visual analog scale, nausea-vomiting and retching index, and mental well-being scales will be applied to all groups at the beginning of the study and three days after the study.

DETAILED DESCRIPTION:
Large Intestine Meridian 4th point (Hegu/LI4), Pericardium Meridian/Neiguan (P6) point and Yintang (EX-HN 3) point will be used for acupressure application in the research.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Cancer patients without distant metastases in stage-1, stage-2 and stage-3 who have received at least one course of chemotherapy
* Pain degree 4 and above (will be evaluated with a visual analog scale)
* Nausea-vomiting degree of 4 and above (will be evaluated with a visual analog scale)
* Receiving standard antiemetic and standard analgesic treatment (All patients included in the study should receive similar treatment.)
* No previous acupressure experience
* Absence of any wound or lesion in the area where acupressure will be applied.
* Not using a different complementary approach during the collection of research data
* Those who signed the Informed Consent Form/Written Consent Form
* Patients without any psychiatric diagnosis will be included in the study.

Exclusion Criteria:

* < 18 years old
* Those who have not received chemotherapy before
* Pain grade below 4 (will be evaluated with a visual analog scale)
* Nausea-vomiting degree below 4 (will be evaluated with a visual analog scale)
* Receiving different antiemetic and analgesic treatments
* Previous acupressure experience
* Any wound or lesion in the area where acupressure will be applied
* Using a complementary approach other than acupressure at the time research data was collected
* Those who did not sign the Informed Consent Form/Written Consent Form
* Patients with any psychiatric diagnosis will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2023-06-05 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-08-24 (Estimated)

PRIMARY OUTCOMES:
Pain intensity will be evaluated with a visual analog scale. | Change from baseline pain level at 3 days
  The patient evaluates their own pain using a scale ranging from 1 to 10, with 1 = very mild discomfort and 10 = the most severe pain the patient can imagine. Ranges for pain intensity; <3 mild pain, 3-6 moderate pain, >6 severe pain.
Nausea-vomiting severity will be evaluated with the Rhodes Nausea-Vomiting and Retching Index. | Change from baseline nausea-vomiting level at 3 days
  Each response is scored as 0 = least distress, 4 = most distress. The patient's experience of nausea and vomiting in each of the 8 items is summed up. The highest possible value is 32, indicating the most severe symptom occurrence score.
Mental well-being will be evaluated using the Warwick-Edinburgh Mental Well-Being Scale. | Change from baseline mental well-being level at 3 days
  The scale is in the 5-point Likert type and a minimum of 14 and a maximum of 70 points are obtained from the scale. Scoring of the scale is (1 = strongly disagree, 2 = disagree, 3 = somewhat agree, 4 = agree, 5 = completely agree).

CONTACTS AND LOCATIONS:
Overall Officials: Esra Çavuşoğlu, Doctorate, Study Director — Mersin University; Hilal Altundal Duru, Doctorate, Principal Investigator — Çankırı Karatekin University; Kadir Eser, Principal Investigator — Mersin University; Emel Sezer, Principal Investigator — Mersin University; Vehbi Erçolak, Principal Investigator — Mersin University; Ümmügülsüm Kılıç, Principal Investigator — Mersin University

IPD SHARING:
Plan to Share IPD: No